CLINICAL TRIAL: NCT07256067
Title: The Effect of Vagus Nerve Acupoint Transcutaneous Electrical Nerve Stimulation on Fatigue in Patients With Systemic Lupus Erythematosus: A Randomized Controlled Trial
Brief Title: Vagus Nerve Stimulation for Fatigue in Systemic Lupus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Asmaa Saed Mahmoud Ebrahim, Teaching assistant in the Department of Surgery and Burns, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2062021
Record Dates: First submitted 2025-09-29; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: System Lupus Erythematosus
Keywords: Vagus Nerve Stimulation; Fatigue; Lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental:Transcutanousvagus nerve stimulation plus aerobic exercise (Experimental): Transcutaneous vagus nerve stimulation (tVNS), combined with aerobic exercise. Stimulation will be applied to the left auricular concha for 20 minutes per session, three times per week for six weeks, using standardized settings (30 Hz frequency, 300 μs pulse width) at a tolerable, non-painful intensity. This will be followed by 40 minutes of aerobic exercises.
  Interventions: Device: transcutaneous vagus nerve stimulation (tVNS)
- sham transcutaneous vagus nerve stimulation (tVNS) plus aerobic exercise (Sham Comparator): sham transcutaneous vagus nerve stimulation (tVNS) using the same device and electrode placement. They will also perform the same 40-minute aerobic exercise program.
  Interventions: Other: sham transcutaneous vagus nerve stimulation (tVNS) plus aerobic exercise

INTERVENTIONS:
Device: transcutaneous vagus nerve stimulation (tVNS) — Transcutaneous auricular vagus nerve stimulation (taVNS) was administered exclusively with fixed stimulation parameters set at a frequency of 30 Hz and a pulse width of 300 μs.3times a week for 6 week.
  * Only spring-loaded clip electrodes were used for stimulation on the left ear.
  * an aerobic exercises designed to improve mobility, strength, and fatigue tolerance lasted 40 minutes and included treadmill, walking andcycling with moderate intensity (60-70% max HR and frequency 3 sessions per week
  * No additional therapies (e.g., resistance training, aquatic therapy, or medications) were included in the intervention.
  Arms: Experimental:Transcutanousvagus nerve stimulation plus aerobic exercise
Other: sham transcutaneous vagus nerve stimulation (tVNS) plus aerobic exercise — sham transcutaneous vagus nerve stimulation (tVNS) using the same device and electrode placement. They will also perform the same 40-minute aerobic exercise program.
  Arms: sham transcutaneous vagus nerve stimulation (tVNS) plus aerobic exercise

SUMMARY:
50female patients diagnosed with systemic lupus erythematosus according to the 2010 Revised American College of Rheumatology (ACR). Their age will range from 35 to 55 years. The participants will be selected from one major healthcare institutions: Al Kaser Al Ayni Teaching hospital, will be randomly equally distributed into two groups.

Group A :(Treatment Group):

This group includes 25 patients diagnosed with systemic lupus erythematosus according to the 2010 Revised American College of Rheumatology (ACR),and will receive transcutaneous vagus nerve stimulation (tVNS), combined with aerobic exercise alongside medical treatment. Patients will receive 3 sessions per week for 6 weeks, the time of session is 45 - 60 min according to patient ability.

Group B :( Control Group) This group includes 25 patients diagnosed with systemic lupus erythematosus according to the 2010 Revised American College of Rheumatology (ACR)and will receive sham transcutaneous vagus nerve stimulation (tVNS) using the same device and electrode placement. They will also perform the same 40-minute aerobic exercise program alongside medical treatment. Patients will receive 3 sessions per week for 6 weeks.

DETAILED DESCRIPTION:
1)Subjects: 50female patients diagnosed with systemic lupus erythematosus according to the 2010 Revised American College of Rheumatology (ACR). Their age will range from 35 to 55 years. The participants will be selected from one major healthcare institutions: Al Kaser Al Ayni Teaching hospital, will be randomly equally distributed into two groups.

Group A :(Treatment Group):

This group includes 25 patients diagnosed with systemic lupus erythematosus according to the 2010 Revised American College of Rheumatology (ACR),and will receive transcutaneous vagus nerve stimulation (tVNS), combined with aerobic exercise alongside medical treatment. Patients will receive 3 sessions per week for 6 weeks, the time of session is 45 - 60 min according to patient ability.

Group B :( Control Group) This group includes 25 patients diagnosed with systemic lupus erythematosus according to the 2010 Revised American College of Rheumatology (ACR)and will receive sham transcutaneous vagus nerve stimulation (tVNS) using the same device and electrode placement. They will also perform the same 40-minute aerobic exercise program alongside medical treatment. Patients will receive 3 sessions per week for 6 weeks.

2)Equipment:

• Therapeutic Equipment: .Transcutaneous auricular vagus nerve stimulation (taVNS) was administered exclusively with fixed stimulation parameters set at a frequency of 30 Hz and a pulse width of 300 μs.

* Only spring-loaded clip electrodes were used for stimulation on the left ear.
* an aerobic exercises designed to improve mobility, strength, and fatigue tolerance lasted 40 minutes and included treadmill, walking andcycling with moderate intensity (60-70% max HR and frequency 3 sessions per week
* No additional therapies (e.g., resistance training, aquatic therapy, or medications) were included in the intervention.

Measurement equipment:

• Fatigue severity scale: is a widely used self-report questionnaire designed to assess the impact of fatigue on daily functioning. It consists of nine statements rated on a 7-point Likert scale, with higher scores indicating greater fatigue severity. The FSS has demonstrated strong psychometric properties in patients with systemic lupus erythematosus (SLE), including excellent internal consistency (Cronbach's α > 0.90) and good test-retest reliability (ICC = 0.84-0.89). The Arabic version of the FSS has been validated in multiple studies and has shown comparable reliability and construct validity to the original version. For example, Al-Sobayel et al. (2016) reported a Cronbach's α of 0.93 for the Arabic FSS in a population of Arabic-speaking patients with chronic diseases, including SLE. This makes the Arabic FSS a culturally appropriate and psychometrically sound instrument for assessing fatigue in Arabic-speaking populations.

Six-Minute Walk Test (6MWT) is a sub-maximal exercise test that measures the distance a person can walk as far as possible in six minutes along a flat, hard surface.

It is used to assess functional exercise capacity, endurance, and the integrated global response of many systems: pulmonary and cardiac function, circulation, peripheral circulation, neuromuscular function, The test can show performance fatigability when there is a decline in the individual's walking speed or distance over time (for instance, comparing the first minute of walking vs the last minute.

Borg Rating of Perceived Exertion (RPE) ("Borg Test") is a subjective scale developed by Gunnar Borg, used to gauge how hard someone feels they are working during physical activity. It captures feelings of exertion, breathlessness, muscle fatigue, heart rate

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 35 to 55 years
* Diagnosis of Systemic Lupus Erythematosus (SLE) based on the 2010 Revised American College of Rheumatology (ACR) or SLICC classification criteria.
* Self-reported pain score of ≥4 on a 10 cm Visual Analogue Scale (VAS).
* Receiving stable doses of Disease Modifying Anti-Rheumatic Drugs (DMARDs), biological therapy, and/or prednisone ≤10 mg/day, with no changes in dose within 28 days prior to baseline.
* They have been referred by a rheumatologist.

Exclusion Criteria:

* Diagnosis of fibromyalgia or any other overlapping chronic pain syndrome.
* Use of pacemakers, implantable cardioverter defibrillators (ICDs), or other electronic implants.
* Current pregnancy or breastfeeding.
* History of epilepsy or seizure disorders.

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-10-02 (Actual); Study Completion 2025-11-02 (Actual)

PRIMARY OUTCOMES:
Fatigue severity scale | 6 weeks
  The Fatigue Severity Scale (FSS) is a widely used self-report questionnaire designed to assess the impact of fatigue on daily functioning. It consists of nine statements rated on a 7-point Likert scale, with higher scores indicating greater fatigue severity. The FSS has demonstrated strong psychometric properties in patients with systemic lupus erythematosus (SLE), including excellent internal consistency (Cronbach's α > 0.90) and good test-retest reliability (ICC = 0.84-0.89). The Arabic version of the FSS has been validated in multiple studies and has shown comparable reliability and construct validity to the original version.

SECONDARY OUTCOMES:
Six-Minute Walk Test (6MWT) andBorg Rating of Perceived Exertion (RPE) (Borg Test) | 6 weeks
  The 6MWT is a sub-maximal exercise test that measures the distance a person can walk as far as possible in six minutes along a flat, hard surface.
  It is used to assess functional exercise capacity, endurance, and the integrated global response of many systems: pulmonary and cardiac function, circulation, peripheral circulation, neuromuscular function, The test can show performance fatigability when there is a decline in the individual's walking speed or distance over time (for instance, comparing the first minute of walking vs the last minute. That was measured by map by walk phone application.
Borg rating scale | 6 weeks
  RPE is a subjective scale developed by Gunnar Borg, used to gauge how hard someone feels they are working during physical activity. It captures feelings of exertion, breathlessness, muscle fatigue, heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Research Ethical Committee, Faculty of Physical Therapy, Principal Investigator — faculty of physical therapy
Locations (1):
- faculty of Physical Therapy, Giza, Egpt, Egypt